CLINICAL TRIAL: NCT02013986
Title: Phase 1 Study of Circadian Rhythm of Salivary Cortisol in Health Children ;Phase 2 Study of Circadian Rhythm of Salivary Cortisol of Children Undergoing Surgery Using Etomidate or Not Using Etomidate.
Brief Title: Effects of Etomidate on Postoperative Circadian Rhythm Changes of Salivary Cortisol in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Du yi (Other)
Responsible Party: Sponsor-Investigator, Du yi, attending of anesthesiology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X01PA131001
Record Dates: First submitted 2013-11-07; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Congenital Hydronephrosis; Congenital Choledochal Cyst; Fracture
Keywords: salivary cortisol; circadian rhythm; children; etomidate
MeSH Terms: conditions — Choledochal Cyst; Fractures, Bone | interventions — Etomidate; Midazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- etomidate & midazolam (Experimental): a bolus of midazolam(Jiangsu Enhua Pharmaceutical Ltd.) 0.1mg/kg then a bolus of etomidate(Etomidate Fat Emulsion Injection, Jiangsu Enhua Pharmaceutical Ltd.)0.3 mg/kg and intravenously, during induction period, the other steps as usual.
  Interventions: Drug: etomidate; Drug: midazolam
- midazolam & propofol (Active Comparator): During induction period,use a bolus of midazolam injection 0.1mg/kg(Jiangsu Enhua Pharmaceutical Ltd.) and then a bolus of propofol injection 2mg/kg(Astrazeneca PLC.)intravenously, the other steps are as usual.
  Interventions: Drug: midazolam; Drug: propofol

INTERVENTIONS:
Drug: etomidate — 0.3mg/kg IV only once during induction of general anesthesia
  Other Names: Fuerli
  Arms: etomidate & midazolam
Drug: midazolam — midazolam 0.1mg/kg IV only once before using of etomidate/propofol during induction of general anesthesia
  Other Names: Liyuexi
Drug: propofol — 2mg/kg IV only once during induction of general anesthesia
  Other Names: Diprivan
  Arms: midazolam & propofol

SUMMARY:
Etomidate is an unique drug used for induction of general anesthesia and sedation. Adrenal cortical inhibition by etomidate has received much attention. However wether the circadian rhythm and pulse secretion pattern of cortisol in children are the same as that in adults is not known. Moreover, the effect of etomidate on circadian rhythm changes and clinical outcomes has never been carefully studied in children undergoing surgery. Our hypothesis is that etomidate can relieve the changes of circadian rhythm of salivary cortisol in children for 24-48 hours，and this does not make clinical outcomes worse postoperatively.

DETAILED DESCRIPTION:
* Sample size assessment: Using formula to calculate the total number is 30.
* Statistical analysis: ANOVA
* Reporting for adverse events: During the period of study, if there is any severe adverse event happening, such as severe infection, severe low cortisol concentration threatening the patient's life we will stop the trial.

ELIGIBILITY:
Inclusion Criteria:

* 3-12 years old who are plan to undergo surgery

Exclusion Criteria:

* endocrine disease, blood infusion, having fever, ulcer or bleeding in the oral cavity

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in salivary cortisol at the operative day | baseline(8am), 8pm
  At the time of 8am(baseline) and at the time of 8pm in the operative day , get salivary samples to calculate the change of salivary cortisol
Change from baseline in salivary cortisol at the first day after surgery | baseline(8am), 8pm
  At the time of 8am(baseline) and at the time of 8pm in the first day after surgery , get salivary samples to calculate the change of salivary cortisol

SECONDARY OUTCOMES:
Numbers of Acquired Infection Events | up to 10 days after surgery
  Acquired infection using extra antibiotics(not prophylactic antibiotics) after surgery.
Numbers of using inotropic drugs | within 3 days
  Inotropic drugs include norepinephrine, adrenaline, phenylephrine and dopamine.
Days of stay in intensive care unit (ICU) after surgery | up to 10 days after surgery
  Days of stay in ICU after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Wng Y Wei, professor, Study Director — Shanghai Jiao Tong University School of Medicine
Locations (1):
- department of anesthesia of Xinhua Hospital, Shanghai, Shanghai Municipality, China